CLINICAL TRIAL: NCT02740309
Title: Integrated Behavioral Health Innovations in Childhood Chronic Illness Care Delivery Systems
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-01065
Record Dates: First submitted 2016-02-24; First posted 2016-04-15 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; childhood chronic disease; adolescent depression; adolescent anxiety; integrated brief behavioral therapy; adolescent psychosocial risks; adolescent chronic disease; childhood depression; childhood anxiety; childhood psychosocial risks
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Methods; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Brief Behavior Therapy (IBBT) Intervention (Experimental): 4-sessions of IBBT for youth anxiety and depression.
  Interventions: Behavioral: Integrated Brief Behavior Therapy (IBBT) Intervention
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Integrated Brief Behavior Therapy (IBBT) Intervention — The 4 sessions will empower and support families and youth to continue treatment autonomously with home practice
  Arms: Integrated Brief Behavior Therapy (IBBT) Intervention
Behavioral: Treatment as usual — Facilitated community referral for mental health treatment
  Arms: Treatment as usual

SUMMARY:
Study design: At baseline, all adolescents and young adults with IBD ages 12-21 years will be screened for anxiety and depression symptoms using the PHQ-9 and the Screen for Child Anxiety Related Disorders (SCARED) during a routine medical visit in the pediatric gastroenterology clinic. Individuals who screen positive for depression or anxiety will be assessed to confirm diagnoses using the anxiety and M.I.N.I. 6.0. Participants will also complete a psychosocial risk assessment as well as medical and socio-demographic inventories. The investigators will include youth that meet full criteria for major depressive disorder and any anxiety disorder, dysthymic disorder, and any adjustment disorder. The investigators will also include patients with subclinical symptoms that have significant psychosocial stressors in addition to their medical illness. Patients will be excluded if they have active suicidal ideation with plan requiring ER referral, bipolar disorder, psychosis, substance dependence, eating disorders, or significant intellectual disability/developmental delay. Participants meeting inclusion criteria will be randomly assigned to four sessions of IBBT administered on-site by a Fink social worker or treatment as usual (TAU), which is a facilitated community referral for mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adolescents and young adults with IBD ages 12-21 years will be screened for anxiety and depression symptoms and includes youth that meet full criteria for major depressive disorder and any anxiety disorder, dysthymic disorder, and any adjustment disorder. The investigators will also include patients with subclinical symptoms that have significant psychosocial stressors in addition to their medical illness.

Exclusion Criteria:

* Patients will be excluded if they have active suicidal ideation with plan requiring ER referral, bipolar disorder, psychosis, substance dependence, eating disorders, or significant intellectual disability/developmental delay.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety and/or Depression Symptoms | 1 year ( baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  Anxiety and depression symptoms are hypothesized to decrease more in the IBBT-4 group and psychosocial functioning is hypothesized to improve more in the IBBT-4 group as compared to TAU. The number of patients who no longer meet criteria for depression and/or anxiety after brief intervention is hypothesized to be greater than as compared to TAU. The Patient Health Questionnaire (PHQ-9) will be repeated self-report measures of depression and anxiety symptoms at each time point to assess symptomatology.The PHQ-9 consists of 9 questions scored 0-3, with 3 denoting the early every day ( highest value).
Treatment Engagement at Baseline | 1 year
  One visit is the modal number of encounters for patients seeking treatment in the community mental health care settings. The investigators hypothesize that by implementing an integrated behavioral health model that identifies mental health issues in medical settings as part of routine care and engages individuals in on-site treatment for depression and anxiety will increase the number of completed mental health encounters utilized and the number of successful referrals to community mental health providers when ongoing treatment is needed.
  Multiple measurements will be aggregated to arrive at 1 reported value.Data will be collected by tracking the number of sessions attended for IBBT-4 vs. the number of sessions attended for the treatment as usual group at 8 weeks post initial assessment as well as whether or not referrals to community mental health providers are successfully completed by either group at each time point.
Screen for Childhood Anxiety Related Emotional Disorders (SCARED) | 1 year
  The SCARED will be repeated self-report measures of anxiety symptoms at each time point to assess symptomatology. SCARED is a 41-item screening tool with each scored from 0 to 2, with 2 denoting "very true or often true" (highest value). Total scores of 25 or greater indicate the presence of an Anxiety Disorder. Subscore cut off ranges are also provided for Panic Disorder or Significant Somatic Symptoms, Generalized Anxiety Disorder, Separation Anxiety, Social Anxiety, and School Avoidance.
Children's Global Assessment Scale (CGAS) | 1 year
  A Children's Global Assessment Scale (CGAS) will also be completed at baseline and at each time point for global psychosocial functioning.C-GAS is rated from 0 to 100, where 1 represents the most impaired functioning and 100 represents superior functioning.
Columbia Suicide Severity Rating Scale (C-SSRS) | 1 year
  At baseline screening, the Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess for suicidal ideation or actions.CSSRS consists of ten categories and have binary responses (yes/no). A "yes" answer at any time during treatment to Categories 1-5 is defined as suicidal ideation. A "yes" answer at any time during treatment to Categories 6-10 is defined as suicidal behavior. A "yes" answer to any one of the ten suicidal ideation and behavior questions at any time during treatment to (Categories 1-10) is defined as suicidal ideation or behavior.

SECONDARY OUTCOMES:
IBD disease activity - Pediatric Ulcerative Colitis Activity Index (PUCAI) | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  IBD disease activity will be assessed through validated Pediatric Ulcerative Colitis Activity Index (PUCAI) which measure symptom severity in a given time period through physician, laboratory, and subjective self-report markers of disease activity. These measures will be assessed at each time point. PUCAI score ranges from 0 to 85; a score of < 10 denotes remission, 10-34 indicates mild disease, 35-64 indicates moderate disease, and 65-85 indicates severe disease.
IBD-related quality of life-SIBDQ | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  IBD-related quality of life will be measured by the Short Quality of Life Questionnaire for Inflammatory Bowel Disease (SIBDQ).
Medical Adherence Measure | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  Medical Treatment Adherence will be measured by the Medical Adherence Measure (MAM).
Health Care Utilization | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  Health care utilization will be measured by outpatient and emergency room visits and inpatient hospitalizations collected through medical record review and participant self-report.
Pediatric Crohn's Disease Activity Index (PCDAI) | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  IBD disease activity will be assessed through validated Pediatric Crohn's Disease Activity Index (PCDAI) which measure symptom severity in a given time period through physician, laboratory, and subjective self-report markers of disease activity.The PCDAI has hematocrit, Albumin and ESR as markers:ESR: 0-20 mm/hr, Albumin: 3.5 - 5.0 gm/dL, HCT: 35-47%. As for the disease indicators: PCDAI score can range from 0-100, with higher scores signifying more active disease. A score of < 10 is consistent with inactive disease, 11-30 indicates mild disease, and > 30 is moderate-to-severe disease.
Health Care Cost | 1 year ( Data will be collected at 4 time points: baseline, 8-12 weeks, 6 months, and 12 months post baseline)
  Health Care costs will be measured by outpatient and emergency room visits and inpatient hospitalizations collected through medical record review and participant self-report.

CONTACTS AND LOCATIONS:
Overall Officials: K. Ron-Li Liaw, MD, Principal Investigator — NYU Langone
Locations (1):
- Sala Institute for Child and Family Centered Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Sala Institute for Child & Family Centered Care: Sala Institute — http://nyulangone.org/locations/hassenfeld-childrens-hospital/sala-institute-for-child-family-centered-care